CLINICAL TRIAL: NCT04475406
Title: Comparison of Bone Immunological Biomarkers and Microbiological Parameters of Extra Short Dental Implants and Standard Dental Implants Loaded in the Posterior Mandible
Brief Title: Comparison of Short and Standard Dental Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Bilge Karcı, Assistant Professor, Alanya Alaaddin Keykubat University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2016/009
Record Dates: First submitted 2020-07-09; First posted 2020-07-17 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Peri-Implantitis; Peri-implant Mucositis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): Standard implant, intra-bone length ≥8 mm (30 implants)
  Interventions: Other: PICF (Periopaper); Other: Subgingival plaque, Gracey curette (Hu-Friedy); Other: Clinical data, williams probe PCPNU (Hu-Friedy)
- Test group (Active Comparator): Extra Short implant, intra-bone length ≤6 mm (30 implants)
  Interventions: Other: PICF (Periopaper); Other: Subgingival plaque, Gracey curette (Hu-Friedy); Other: Clinical data, williams probe PCPNU (Hu-Friedy)

INTERVENTIONS:
Other: PICF (Periopaper) — After the plaques and soft attachments around the implants were removed, the implants were isolated using cotton rolls and dried with an air spray. The PICF was collected from the mesio-buccal region of the implant using periopaper strips (Oraflow Inc, NY, USA). Paper strips were placed 1-2 mm inside the peri-implant sulcus and kept for 30 s. Paper strips were placed in sterile Eppendorf tubes containing 200 µL of phosphate-buffered saline (PBS). The tubes were kept at -80°C until the analysis day. Paper strips contaminated with saliva or blood were excluded from the sampling.
Other: Subgingival plaque, Gracey curette (Hu-Friedy) — After collecting the PICF, the supragingival plaque was carefully removed using a sterile scaler. Implants were isolated using cotton rolls and dried with an air spray. Subgingival plaque samples were collected from the mesio-buccal region of the implant using a sterile plastic Gracey curette (Hu-Friedy, Switzerland) for 30 s. The samples collected were transferred to sterile Eppendorf tubes containing 200 µL of PBS. The tubes were kept at -80°C until the analysis day.
Other: Clinical data, williams probe PCPNU (Hu-Friedy) — A single calibrated examiner performed all (full-mouth and site-specific) clinical measurements (B.K.), including probing depth (PD), clinical attachment level (CAL), presence of bleeding on probing (BOP), 3-year survival rate (CSR), and bone loss (BL).
  The values of PD and BOP were measured from four sites of each implant (mesial, distal, buccal, and lingual) with a Williams type (Hue Friedy, Switzerland) plastic periodontal probe. The PD was recorded as the distance from the base of the peri-implant to the side of the gum in millimeters. BOP was evaluated according to the presence (+) or absence (-) of bleeding within the first 30 s following the measurement of PD.17 Control panoramic films of all patients were taken, and differences in the marginal bone level between radiography images after implant placement and 3 years later were evaluated. Original films and images taken later were taken with the same angle for standardizaton.

SUMMARY:
Objective: This study aimed to evaluate the total amounts of tumor necrosis factor α (TNF-α), prostaglandin E2 (PGE2), receptor activator of nuclear factor kappa B ligand (RANKL), receptor activator of nuclear factor kappa B (RANK), and osteoprotegerin (OPG) and the abundance of putative oral pathogens Fusobacterium nucleatum, Porphyromonas gingivalis, Treponema denticola, Tannerella forsythia, Prevotella intermedia, and Streptococcus oralis in extra short and standard dental implants functioning in the posterior mandible.

Methodology: The implants were divided into two groups according to their lengths: standard (intrabony length ≥8 mm) and extra short (intrabony length ≤ 6 mm). A total of 60 implants were researched in 30 patients. Probing depth (PD), clinical attachment level (CAL), presence of bleeding on probing (BOP), 3-year survival rate (CSR), and bone loss (BL) were measured.

DETAILED DESCRIPTION:
INTRODUCTION

Dental implants are usually considered an alternative treatment option to replace lost teeth in edentulous patients. The rate of implant placement in regions more difficult to rehabilitate has increased with the increase in the success of osseointegration and survival. However, besides implant placement in sites with insufficient crest width and height, treatment times and costs have also increased with the use of grafting procedures.1 Various surgical techniques, such as vertical bone augmentation, sinus floor elevation, and nerve transposition, have been developed for the treatment of these bone volume insufficiencies. However, these methods are technically sensitive and can cause significant postoperative complications. Short dental implants have been suggested as a simpler, cheaper, and faster alternative to prevent the disadvantages of surgical techniques and for the rehabilitation of toothless areas.2,3 A large number of randomized controlled clinical trials demonstrated that the long-term success and survival rates of short implants were similar to those of standard long implants.4-6 Accumulation of microbial dental plaque around the implant is the most important cause of implant loss. If the microbial attachment is not removed, diseases such as peri-implant mucositis and peri-implantitis may occur and result in implant loss in the long term. Peri-implant mucositis is a reversible inflammatory reaction in the soft tissue surrounding the implant in function. Peri-implantitis is a microbial inflammatory disease characterized by the resorption of the supportive bone surrounding the implant in function.7 Gram-negative anaerobic bacteria predominate around the implant sites affected by the disease. While they resemble chronic periodontal infections, they have a more complex microbiological character.8 Predominant species around a peri-implantitis implant are red complex (P. gingivalis, T. denticola, and T. forsythia) and orange complex bacteria (F. nucleatum and P. intermedia) described by Socransky.9 In 1989, Apse et al. reported a fluid around the peri-implant sulcus with properties similar to those of the gingival crevicular fluid, and they called this fluid peri-implant crevicular fluid (PICF).10 The PICF is an inflammatory exudate formed by osmotic pressure. Biochemical mediators in the PICF are highly important to determine the health of tissues around the implant.11 Prostaglandins, especially prostaglandin E2 (PGE2), are considered as a potent mediator of alveolar bone destruction in periodontitis. A large number of studies reported an increase in PGE2 levels from healthy state to periodontitis.12 Tumor necrosis factor α (TNF-α) is a proinflammatory cytokine regulating the Gram-negative bacterial response. The TNF-α concentration is an indicator of bacterial load and degree of inflammation.13 In areas where peri-implantitis is active, the presence and activity of osteoclasts are necessary for bone destruction to occur. The formation and activation of osteoclasts are regulated through the activation of three members of the TNF family: receptor activator of nuclear factor kappa B ligand (RANKL), receptor activator of nuclear factor kappa B (RANK), and osteoprotegerin (OPG). Osteoclast differentiation and activation occur with the binding of RANKL to RANK over the surface of osteoclasts and precursors. OPG, which is a soluble protein of TNF receptors, antagonizes RANK-RANKL interaction and increases bone formation by inhibiting osteoclastogenesis. The levels of proinflammatory cytokines, such as IL-1, IL-6, TNF-α, and PGE2, and RANKL/OPG rates, which allow the determination of osteoclastic activity, change in the case of peri-implantitis.14 The aim of this study was to evaluate the levels of TNF-α, PGE2, RANKL, RANK, and OPG in extra short and standard dental implants functioning in the posterior mandible. An additional aim was to investigate the levels of putative oral pathogens F. nucleatum, P. gingivalis, T. denticola, T. forsythia, P. intermedia, and S. oralis in submucosal biofilm samples from the studied sites.

MATERIALS AND METHODS This study was carried out by recalling individuals whose bilateral partial tooth losses were treated with implant-supported fixed restorations and whose implants had been functioning for at least 3 years after prosthetic rehabilitation. The study was conducted in accordance with the ethical guidelines from the World Medical Association Declaration of Helsinki (version 2013) (Clinical Researches Ethical Board with the 28. 09. 2016 and 2016/009 decision numbered approval).

A total of 31 patients met the inclusion criteria. One patient did not continue the study. Further, 60 implants were researched in 30 patients (16 female and 14 male). The bilateral regions of patients with a standard implant and an extra short implant were grouped into two.16 Control group: Standard implant, intra-bone length ≥8 mm (30 implants) Test group: Extra Short implant, intra-bone length ≤6 mm (30 implants)

Collection of clinical data A single calibrated examiner performed all (full-mouth and site-specific) clinical measurements (B.K.), including probing depth (PD), clinical attachment level (CAL), presence of bleeding on probing (BOP), 3-year survival rate (CSR), and bone loss (BL).

The values of PD and BOP were measured from four sites of each implant (mesial, distal, buccal, and lingual) with a Williams type (Hue Friedy, Switzerland) plastic periodontal probe. The PD was recorded as the distance from the base of the peri-implant to the side of the gum in millimeters. BOP was evaluated according to the presence (+) or absence (-) of bleeding within the first 30 s following the measurement of PD.17 Control panoramic films of all patients were taken, and differences in the marginal bone level between radiography images after implant placement and 3 years later were evaluated. Original films and images taken later were taken with the same angle for standardizaton.

Collection of PICF and subgingival plaque samples After the plaques and soft attachments around the implants were removed, the implants were isolated using cotton rolls and dried with an air spray. The PICF was collected from the mesio-buccal region of the implant using periopaper strips (Oraflow Inc, NY, USA). Paper strips were placed 1-2 mm inside the peri-implant sulcus and kept for 30 s. Paper strips were placed in sterile Eppendorf tubes containing 200 µL of phosphate-buffered saline (PBS). The tubes were kept at -80°C until the analysis day. Paper strips contaminated with saliva or blood were excluded from the sampling.

After collecting the PICF,. the supragingival plaque was carefully removed using a sterile scaler. Implants were isolated using cotton rolls and dried with an air spray. Subgingival plaque samples were collected from the mesio-buccal region of the implant using a sterile plastic Gracey curette (Hu-Friedy, Switzerland) for 30 s. The samples collected were transferred to sterile Eppendorf tubes containing 200 µL of PBS. The tubes were kept at -80°C until the analysis day.

PICF analysis Commercial enzyme-linked immunosorbent assay kits were used for measuring the levels of TNF-α, PGE2, RANKL, RANK, and OPG in accordance with the manufacturer's recommendations (Elabscience Biotechnology Co., Ltd, Wuhan, China). The measuring ranges were as follows: TNF-α, 7.81-500 pg/mL; PGE2, 31.25-2000 pg/mL; RANKL, 0.16-10 pg/mL; RANK, 0.16-10 pg/mL; and OPG, 0.16-10 pg/mL. Optical density was measured at 450 nm, and the samples were compared with standards. Biochemical data were measured as the total amount (pg/30 s).

Genomic DNA preparation An extraction kit was used in accordance with the manufacturer's recommendations to purify the DNA in the collected plaque samples (GF-1 bacterial DNA extraction kit, Vivantis, Malaysia). Standards were used for total DNA in the target bacteria. Genomic DNA was obtained and stored at 4°C.

Real-time polymerase chain reaction Primary probes were determined to define each bacterium and observe the proliferation curves using real-time polymerase chain reaction (PCR) (Table 1). For the DNA amplification reaction, procedures were performed with a real-time PCR system (Roche Light Cycler 480 Instrument II, Switzerland) using a master mix (SYBR Green Master Mix; Life Technologies, CA, USA). PCR cycles were as follows: 10 min at 95°C, 40 cycles at 95°C for 30 s and 2 min at 60°C. DNA contents were calculated using standard curves.

Statistical analysis Statistical analyses were performed with SPSS 19.0 (IBM Inc., IL, USA). Kolmogorov-Smirnov and Shapiro-Wilk tests were used to examine whether the variables were normally distributed. The level of significance was used as 0.05 while commenting on the results.

While examining the differences between the groups, the independent-samples t test was used when the variables were normally distributed.

The nonparametric Mann-Whitney U test was used when the variables were not normally distributed. The chi-square analysis was used while examining the relationships between the groups of nominal variables. The survival rate (CSR) was calculated according to the number of short and standard implants placed.

ELIGIBILITY:
Inclusion Criteria:

* Implants placed by the same periodontologist (E.Ö.) functioning for at least 3 years
* Patients without any systemic disease affecting bone metabolism
* Age >18 years
* Extra short (6-mm) implants with identical surface properties bilaterally in one area in the mandibular region and standard (≥8 mm) implants in the other area
* Placed implants having the same brand (Straumann Standard Plus; Institute Straumann AG, Basel, Switzerland)
* Patients with cemented implant prosthesis in which standard abutment was used in the mandibular posterior region
* Implants having no additional bone augmentation during implant surgery
* No periodontal treatment received in the last 3 years
* Patients under oral hygiene control (plaque score <20%)

Exclusion Criteria:

* Poor oral hygiene (plaque score >20%)
* Patients with a history of periodontitis
* Uncontrolled diabetes and other uncontrolled diseases
* Pregnancy and lactation
* Smoking more than 10 cigarettes a day
* Using alcohol
* Receiving radiotherapy and chemotherapy
* Using drugs suppressing the immune system
* Having a parafunctional habit

Ages: 35 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
the levels of putative oral pathogens (using PCR) | an average of 3 year
  An extraction kit was used in accordance with the manufacturer's recommendations to purify the DNA in the collected plaque samples (GF-1 bacterial DNA extraction kit, Vivantis, Malaysia). Standards were used for total DNA in the target bacteria. Primary probes were determined to define each bacterium and observe the proliferation curves using real-time polymerase chain reaction (PCR)

SECONDARY OUTCOMES:
total amount of TNF-α, PGE2, RANKL, RANK, and OPG (using ELISA) | an average of 3 year
  Commercial enzyme-linked immunosorbent assay kits were used for measuring the levels of TNF-α, PGE2, RANKL, RANK, and OPG in accordance with the manufacturer's recommendations (Elabscience Biotechnology Co., Ltd, Wuhan, China).

CONTACTS AND LOCATIONS:
Overall Officials: Bilge Karcı, Dr., Study Director — Alanya Alaaddin Keykubat University

IPD SHARING:
Plan to Share IPD: No
After 1 years